CLINICAL TRIAL: NCT07311395
Title: Local Subcutaneous Administration of Gentamicin for the Prevention of Surgical Site Infection Following Elective Cesarean Section: A Randomized Controlled Pilot Study.
Brief Title: Local Subcutaneous Gentamicin for Prevention of Surgical Site Infection After Elective Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Nadir Ganem, Principal Investigator, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0177-25-NHR
Record Dates: First submitted 2025-12-15; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Gentamicins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local subcutaneous gentamicin (Experimental)
  Interventions: Drug: Gentamicin
- Standard antibiotc prophylaxis (Active Comparator)
  Interventions: Drug: Standard antibiotic prophylaxis

INTERVENTIONS:
Drug: Gentamicin — Participants receive a single local subcutaneous administration of gentamicin at the surgical site during elective cesarean section, in addition to standard systemic antibiotic prophylaxis, to reduce postoperative surgical site infection.
  Arms: Local subcutaneous gentamicin
Drug: Standard antibiotic prophylaxis — Participants receive standard systemic antibiotic prophylaxis according to institutional protocol.
  Arms: Standard antibiotc prophylaxis

SUMMARY:
The goal of this clinical trial is to evaluate whether local subcutaneous administration of gentamicin reduces the incidence of surgical site infection (SSI) following elective cesarean section. The study will also assess the safety of local gentamicin administration. The main questions this study aims to answer are:

* Does local subcutaneous administration of gentamicin reduce the rate of superficial and deep surgical site infections within 30 days after elective cesarean delivery?
* Are there differences between groups in postoperative complications, including wound healing, fever, need for additional antibiotic treatment, or hospital readmission?

Researchers will compare women who receive local subcutaneous gentamicin at the surgical site in addition to standard antibiotic prophylaxis to women who receive standard antibiotic prophylaxis alone.

Participants will:

* Undergo an elective cesarean section according to standard clinical practice
* Receive either local subcutaneous gentamicin administration or no local antibiotic administration, in addition to standard systemic antibiotic prophylaxis
* Be followed clinically for signs of surgical site infection and other postoperative complications during hospitalization and at follow-up visits up to 30 days after surgery

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older. Undergoing elective cesarean section. Gestational age >= 24 weeks. Planned postoperative follow-up of 30 days. Eligible for standard antibiotic prophylaxis according to institutional protocol.

Able to provide informed consent.

Exclusion Criteria:

* Known allergy of hypersensitivity to aminoglycosides. Known allergy of hypersensitivity to systemic antibiotic prophylaxis agents. Current or planned use of immunomodulatory or immunosuppressive therapy. Requirement for therapeutic ( non- prophylactic) antibiotic treatment at the time of surgery.

Active infection or clinical condition requiring antibiotic treatment. Inability or unwillingness to comply with study procedures or follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is limited to individuals of the female biological sex due to the nature of elective cesarean delivery.
Enrollment: 100 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
postoperative surgical site infection | within 30 days after cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital-Nahariya, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No